CLINICAL TRIAL: NCT01024543
Title: Role of Angiotensin II in Insulin-induced Microvascular Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. CDA Stehouwer, Maastricht University Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 06-2-074
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Insulin Sensitivity; Microcirculation
Keywords: Angiotensin II
MeSH Terms: conditions — Insulin Resistance | interventions — Angiotensin II; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Sham Comparator): Placebo
  Interventions: Drug: Placebo
- Angiotensin II (Experimental): Angiotensin II
  Interventions: Drug: Angiotensin II
- Phenylephrine (Active Comparator): Phenylephrine
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II
  Arms: Angiotensin II
Drug: Phenylephrine — Phenylephrine
  Arms: Phenylephrine
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study we hypothesize infusion of Angiotensin II improves the insulin-induced microvascular dilatation and therefore insulin-mediated glucose uptake. Objectives: Does infusion of Angiotensin II increase insulin-mediated glucose uptake via enhanced insulin-mediated microvascular function in healthy subjects?

ELIGIBILITY:
Inclusion Criteria:

1.18-60 years 2.Caucasian 3.Blood pressure <140/90 mmHg.

Exclusion Criteria:

1. Obesity (BMI>27kg/m2)
2. Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, heart failure)
3. Impaired glucose tolerance or diabetes mellitus according to the criteria of the ADA
4. Smoking
5. Alcohol use >4U/day
6. Use of medication (antihypertensive drugs, lipid lowering drugs, corticosteroids, NNSAIDs)
7. Pregnancy
8. Wearing contact lenses

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11

PRIMARY OUTCOMES:
functional recruitment of capillaries in the skin | January 2009

SECONDARY OUTCOMES:
perfused capillary density in the nailfold | January 2009
Endothelium- (in)dependent vasodilatation of finger skin microcirculation | January 2006
Insulin sensitivity | January 2009

CONTACTS AND LOCATIONS:
Overall Officials: CDA Stehouwer, Prof, Study Chair — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, P.o. Box 5800, Netherlands, Netherlands